CLINICAL TRIAL: NCT02871245
Title: Clinical Trial on Acupuncture Therapy in Patients With Gastrointestinal Neoplasms Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaonan Cui (Other)
Responsible Party: Sponsor-Investigator, Xiaonan Cui, Professor, Chief physician, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2016-38
Record Dates: First submitted 2016-08-07; First posted 2016-08-18 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Acupuncture Therapy; Laparoscopic Surgery; Gastrointestinal Tract Recovery of Function
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Laparoscopy; Acupuncture Therapy

ARMS (2):
- Comparator Group (Active Comparator): Patients received gastrointestinal neoplasms laparoscopic surgery but no acupuncture therapy.
  Interventions: Procedure: Laparoscopic Surgery
- Acupuncture Therapy Group (Experimental): Patients received gastrointestinal neoplasms laparoscopic surgery and acupuncture therapy. Finish surgery up to 24 hours electricity acupuncture treatment, treatment 1 times a day, every time lasted 30 minutes, 5 days in a row
  Interventions: Procedure: Laparoscopic Surgery; Device: Acupuncture treatment

INTERVENTIONS:
Procedure: Laparoscopic Surgery
Device: Acupuncture treatment
  Arms: Acupuncture Therapy Group

SUMMARY:
Patients accepted laparoscopic radical operation for carcinoma of colon and upper middle section of the rectum will be as the research object. Cancer patients are diagnosed based on pathology or cell biology. The trial is randomized, parallel and open. They are randomized into 2 groups: both groups receive surgery. The experimental group receives conventional treatment combine with electroacupuncture Zusanli point .etc finish operation and the contrast receives the same conventional treatment with experimental group. Clinical evaluation includes gastrointestinal tract recovery of function, pain relief, life quality improvement. Blood biochemistry tests mainly include gastrin(GAS), stress related hormone, peroxidatic reaction and the ratio of immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Weight: 40kg-90kg, male and female.
* Diagnosis: imaging, cell and pathology report.
* Brain, heart, lung, liver, kidney are at good condition in 2 weeks before surgery.
* No conscious obstacle and limbs disability.

Exclusion Criteria:

* Fainting during acupuncture.
* Electrolyte imbalance.
* Serious and life-threatening complications after surgery.
* In addition, patients taking part in other clinical trials, being treated with other biotherapy or immunotherapy and researchers consider not suitable for clinical subjects for other reasons will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants and classification with operation-related adverse events as assessed by CTCAE v4.03. | day 1, day 3, day 5, day 7 after surgery

SECONDARY OUTCOMES:
The quality of life questionnaire(QLQ). | day 1, day 3, day 5, day 7 after surgery
  Assessing in 5 grade, mainly include appetite, sleep, pain,etc.
Stress hormone in blood. | day 2, day 7 after surgery
  Estradiol (female), progesterone (female), testosterone (male)
Immune cell number ratio in blood. | day 2, day 7 after surgery
  Th1/Th2, Th17/Treg

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD, PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided